CLINICAL TRIAL: NCT03341572
Title: The Effect of Positive End Expiratory Pressure on Central Venous Pressure Among Patients With Different Lung Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jingyuan,Xu (Other)
Responsible Party: Sponsor-Investigator, Jingyuan,Xu, Attending doctor, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017ZDSYLL094-P01
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Sepsis; ARDS; Traumatic Brain Injury
MeSH Terms: conditions — Sepsis; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high response group (Experimental): patients undergo 5,10 and 15cmH2O positive end expiratory pressure ,the change of central venous pressure is more than 2.5cmH2O
  Interventions: Other: 5,10 and 15cmH2O positive end expiratory pressure
- low response group (Placebo Comparator): the change of CVP is less than 2.5cmH2O
  Interventions: Other: 5,10 and 15cmH2O positive end expiratory pressure

INTERVENTIONS:
Other: 5,10 and 15cmH2O positive end expiratory pressure — every patients undergo 5,10 and 15cmH2O positive end expiratory pressure,and observe the central venous pressure of the mentioned points

SUMMARY:
To observe the effect of PEEP on CVP among patients with different respiratory compliance

DETAILED DESCRIPTION:
30 patients with mechanical ventilation and inserted central venous line will be entered. After gathering demographic data, patients undergone 5,10 and 15cmH2O PEEPs and the respective CVPs of the mentioned points will be recorded. According to the change of CVP, the patients will be divided into high response group and low response group, then comparing the lung compliance and thorax elastic resistance differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mechanical ventilation and inserted central venous line

Exclusion Criteria:

1. The age is less than 18 years old or more than 80 years old；
2. Pregnant and lying-in woman；
3. Patients undergoing fluid resuscitation and the speed is more than 200ml/h；
4. Patients with norepinephrine dose are greater than 15 micro per minute；
5. Patients with pericarditis、pulmonary heart disease、right heart failure、atrial fibrillation；
6. Patients with COPD(endogenous PEEP is more than 2cmH2O)、tension pneumonthorax、acute episode asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-13 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
CVP | half an hour
  Measure the central venous pressure of the three level PEEPs of 5,10 and 15cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: yi yang, doctor, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No